CLINICAL TRIAL: NCT02936011
Title: DISsection RE-entry Evaluation With Absorb Bioresorbable Vascular Scaffolds in Chronic Total Occlusion. The DISCRETE CTO Study.
Brief Title: DISsection RE-entry Evaluation With Absorb Bioresorbable Vascular Scaffolds in CTO.
Acronym: DISCRETE-CTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Bristol Royal Infirmary (Unknown); Golden Jubilee National Hospital (Other Government); Royal Infirmary of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15094SW-AS
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CTO PCI with Absorb BVS (Other): Single arm observational after successful CTO PCI with Absorb BVS after antegrade or retrograde dissection and re-entry
  Interventions: Device: CTO PCI using Absorb Bioresorbable Vascular Scaffolds

INTERVENTIONS:
Device: CTO PCI using Absorb Bioresorbable Vascular Scaffolds — CTO PCI

SUMMARY:
Percutaneous Coronary Intervention (PCI) is increasingly effective to treat Chronic Total Occlusion (CTO) lesions in coronary arteries. This trial will examine modern dissection and re-entry approaches to treat more complex CTO lesions with the Absorb Bioresorbable Vascular Scaffold (BVS).

DETAILED DESCRIPTION:
This is a pilot study, with the aim of hypothesis generation. This research aims to establish the feasibility and safety of treating chronic total occlusions using dissection and re-entry techniques in combination with everolimus-eluting bioresorbable vascular scaffolds (Absorb BVS).

Primary aims of the study are:

* To demonstrate a low rate of Target Vessel Failure (stent thrombosis, restenosis or late closure) at 12 and 24 months after CTO PCI and stenting with the Absorb BVS
* To demonstrate a high degree of endothelial stent strut coverage at 12 and 24 moths after CTO PCI and stenting with the Absorb BVSThe primary outcome measure is

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient >18 years old with capacity to provide informed consent
* Females of childbearing potential have a negative pregnancy test
* Subject understands the trial requirements, the treatment procedures and provides written informed consent
* Presence of Chronic Total Occlusion (CTO) in a main epicardial coronary vessel that is known or presumed to be of at least 3 months in duration
* The CTO has been crossed using ADR or RDR techniques and subintimal wire passage is documented on IVUS
* Target vessel is >2.5mm and <4mm in diameter and the lesion can the diseased segment can be covered with 3 Absorb BVS stents
* Target lesion is fully prepared and dilatable before BVS insertion • Absorb BVS are successfully implanted in the target lesion

Exclusion Criteria:

* Acute myocardial infarction with ongoing ST-elevation
* Cardiogenic shock
* Left ventricular ejection fraction <20%
* Subject has one of the following (as assessed prior to the index procedure): - Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months; Current problems with substance abuse; There is a planned non-cardiac procedure that may cause non-compliance with the protocol or confound data interpretation
* Subject will has a condition meaning they are unlikely to tolerate dual antiplatelet therapy for 12 months Subject is treated by dialysis or has a baseline serum creatinine level >220 μmol/L (2.5 mg/dL)
* Known allergy to to contrast (that cannot be adequately premedicated) and/or the trial stent system or protocol-required concomitant medications (e.g. Everolimus or PLLA polymer, all P2Y12 inhibitors, or aspirin)
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint OR subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Need for ongoing long-term anticoagulation
* Subject has received an organ transplant or is on a waiting list for an organ transplant •Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months
* Presence of a stent occlusion or the subject was previously treated at any time with intravascular brachytherapy
* Subject has a clinically significant bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure as per ARC criteria (composite occurrence of any revascularization of the target lesion, myocardial infarction (MI) related to the target vessel, or cardiac death) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Walsh, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Belfast Health & Social Care Trust, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No